CLINICAL TRIAL: NCT06258239
Title: Influence of the Communication Between the Nursing Staff and the Patient on the Analgesic Treatment Effectiveness After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0128-22-ZIV
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-03

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel design - subjects are allocated into one of two study arms
Who Masked: Participant, Outcomes Assessor
Masking Description: Nursing staff who will administer the treatment will not be blinded, given that they will receive instructions regarding text to be communicated with participants while administrating the treatment. The participants and the outcomes assessors will not know which study arm they entered (both will be blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced communication (Other): In the enhanced communication study arm the nurse will say to the patient: "I will now give you a combination of two drugs that will greatly ease your pain. One of the two drugs is morphine, which is a drug from the opioid family, which is the strongest drug family for pain relief that medicine has to offer. This drug is very effective against severe pain after surgery. In addition, the second drug is called XEFO. This drug is from the family of non-steroidal anti-inflammatory drugs. We know that the combination of these two drugs is particularly successful in reducing the kind of pain that you experience. According to my experience, you will feel significant pain relief very soon. I will come to you every 10 minutes to assess if you are still in pain. As long as you are suffering from pain, I will continue to give you additional doses of the treatment. We are allowed to give up to 4 doses of treatment. As the treatment is very strong, not everyone needs all 4 doses".
  Interventions: Other: Communication between nursing staff and participants
- Normal communication (Other): In the normal communication study arm the communication between the nurse and patients will be as usual in clinical practice - i.e. - no instruction are given to the nurses regarding on how to communicate with patients while administrating the treatment.
  Interventions: Other: Communication between nursing staff and participants

INTERVENTIONS:
Other: Communication between nursing staff and participants — The analgesic treatment that will be given are part of clinical routine - the participants will get the same exact treatment regardless if they entered the study and to which study arm they entered. The effect that we are interested to capture is the potential added value of communication between the nursing staff and participants while administrating analgesics.

SUMMARY:
Acute pain is a normal response to tissue injury or disease and has an important biological function. It is adaptive and promotes recuperation by restricting behaviors that might incur further tissue trauma. In the case of post-operative acute pain, the cause and time of the physical injury are known, and because the condition is self-limiting it requires only short-term care. However, if acute pain responses cannot be adequately suppressed, cardiac, pulmonary and neuroendocrine functions may be compromised, and the immune system suppressed.

Inadequate management of post-operative acute pain is a major burden for healthcare services and can contribute to medical complications including inflammation of the respiratory tract, damage to the oxygen supply to the heart muscle, deep vein thrombosis, delayed healing as well as the development of chronic pain, more difficult to treat. In addition, suboptimal management of pain after surgery may impair sleep and have negative psychological effects, such as anxiety, fear and lack of sleep. Proper treatment of pain reduces morbidity, damages, treatment costs, improves the patient's quality of life and his chances of a full recovery. It is therefore essential that all patients undergoing surgery should receive adequate pain management.

Despite years of advances in pain management, the mainstay of postoperative pain therapy in many settings is still opioids. Morphine is the most commonly used opioid to treat moderate to severe pain after surgery in the recovery unit. The growing concern about the significant side effects, addictions and costs of opioids as a drug treatment has led to an urgent need to identify other agents and approaches to postoperative pain management that are effective, safe and cheap.

The main purpose of this study is to examine whether the type of communication between the nursing staff and the patient will affect the results of pain relief treatment in the postoperative recovery department. As a secondary objective, we will examine whether personality traits will predict the effectiveness of the treatment.

DETAILED DESCRIPTION:
We will assess whether the communication style between the nursing staff and the patient will affect the effectiveness of the analgesic treatment after surgery. Communication is the independent variable in this study. Two approaches with be used in this study - increased communication and normal communication styles: Increased communication and normal (or standard). In the increased communication study arm the nurse will say to the patient (before administration of first bolus): "I will now give you a combination of two drugs that will greatly ease your pain. One of the two drugs is morphine, which is a drug from the opioid family, which is the strongest drug family for pain relief that medicine has to offer. This drug is very effective against severe pain after surgery. In addition, the second drug is called XEFO. This drug is from the family of non-steroidal anti-inflammatory drugs (NSAIDS). We know that the combination of these two drugs is particularly successful in reducing the kind of pain that you experience. According to my experience, you will feel significant pain relief very soon. I (the nurse) will come to you every 10 minutes to assess if you are still in pain. As long as you are suffering from pain, I will continue to give you additional doses of the treatment. We are allowed to give up to 4 doses of treatment. As the treatment is very strong, not everyone needs all 4 doses". In the normal communication study arm the communication between the nurse and patients will be as usual in clinical practice - i.e. - no instructions are given to the nurses regarding on how to communicate with patients.

All participants in the study, regardless of the study conditions to which they will be placed, will receive exactly the same pain management protocol as it is accepted in the clinical field. The patient's participation in the study will not have any influence on the treatment he will receive. Only patients who reported pain of 7 or more and who can receive the research treatment (blood oxygen level 92% or higher, heart rate over 50) will be included in the data analysis. Since the data analysis will include only cases in which a pain of 7 or more was reported, we will only detail the treatment protocol of these cases. According to the pain relief protocol (Appendix 1) implemented in the recovery department, the patients will receive both opioids and additional treatment, according to the following guidelines: administration of morphine by impulse (I.V), in doses of 3 mg up to a total of 4 doses (12 mg) on demand at 10 minute intervals, and at the same time with each dose additional treatment is given. As long as the patient reports pain higher than 3, we will continue to give impulse doses (up to 4 doses).

In addition to each dose of morphine, a second treatment will be administered according to the following protocol: the patient suffering from pain will usually receive a first dose of morphine and at the same time will receive IV Xefo, which is a drug from the Non-steroidal anti-inflammatory drugs (NSAID) family. At the second pain assessment (about 10 minutes later), if the patient is still suffering from pain, he will receive a second dose of morphine and at the same time IV Optalgin (on the condition that the patient did not receive this drug in the operating room). At the third pain assessment, if the patient is still suffering from pain, he will receive a third dose of morphine and at the same time IV Paracetamol. Finally, at the fourth pain assessment, if the patient reports that he is still suffering from pain, he will receive a fourth dose of morphine alone (without any additional treatment).

The assessment of treatment effectiveness will be based on two key variables: the intensity of the patient's pain and the number of doses of opioids. The nursing staff member will contact the patient at five time points, once every 10 minutes in order to assess his pain. Pain evaluation will be carried out by a verbal scale (NRS, numerical rating scale 0-10). The number of doses of opioids the patient received (ranging from 1 to 4), which represent a total of four different doses (3, 6, 9 or 12 ml), will be noted. We will assess the personality traits and expectation of pain by asking: how severe do you expect your pain to be after surgery on a scale from 0-10? Self-awareness will be assessed using the Self-Consciousness Scale (SCS-R). Empathy of the therapist will be assessed with two questionnaires: Consultation And Relational Empathy measure (CARE) and the Toronto Empathy Questionnaire (TEQ). The general tendency of a person to respond to the suggestions of others will be assessed by the Short Suggestibility Scale questionnaire (SSS) and optimism will be assessed by Life Orientation Test questionnaire (LOT-R). All questionnaires are in both Hebrew and Arabic languages. In addition, we will use physiological indicators that are collected in the clinical routine in the department including: blood pressure, pulse, saturation (blood oxygen level), respiratory rate, body temperature, level of alertness, pain assessment, documentation of painkillers administration, skin integrity assessment, surgical wound assessment.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible to participate to this study, patients have to be able to provide signed and dated written informed consent and to be compliant with the schedule of protocol assessments. Both gender aged 18 till 80, with creatinine levels under 1.4 and undergoing one of following surgery under general anesthesia will be eligible for this study: Gallbladder surgery, hemorrhoid surgery, hernia surgery, nasal septum correction surgery, endoscopic surgery of the sinuses.

Exclusion Criteria:

Patients with creatinine levels above 1.4, weighing less than 50 kg and patients with mental retardation and cognitive impairment will not be enrolled in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 day (At five time points, every 10 minutes)
  A 0-10 VAS scale ranging "no pain" to "worst imaginable pain"
Opioids consumption | 1 day (Up to 4 time points, every 10 minutes)
  Number of doses of opioids requested

CONTACTS AND LOCATIONS:
Overall Officials: Roi Treister, PhD, Principal Investigator — University of Haifa
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon reasonable request